CLINICAL TRIAL: NCT00300339
Title: Double-Blind, Double-Dummy, Randomized, Parallel Group Trial of SL650472 (Three Dose Regimens Versus Placebo and Cilostazol), for 24-Week Improvement of Walking Distance in Patients With Stage II Peripheral Arterial Disease Who Benefit From Optimal Prevention Strategy Including Clopidogrel
Brief Title: Mixed Antagonist of Serotonin for Claudication Optimal Therapy
Acronym: MASCOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT4791
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SL650472, Clopidogrel

SUMMARY:
To investigate in patients suffering from intermittent claudication due to Fontaine stage II PAD whether a 24-week treatment by SL650472 OD on top of clopidogrel may result in an improvement of walking capacity, by comparing three doses of SL650472 to placebo, and to calibrate such effect versus cilostazol

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient with stable symptoms of intermittent claudication of the lower extremities, secondary to chronic occlusive arterial disease from atherosclerosis origin (symptoms present for 6 months or longer and not significantly changed within the past 3 months);
* 2. ICD of 30 to 200 m at screening constant workload treadmill test
* 3. Doppler-measured pre-treadmill ABI of 0.90 or lower after 10 minutes of rest or, for patients with an ABI of greater than 1.3 (non-compressible arteries), a Toe-Brachial Index (TBI) of less than 0.7.

Exclusion Criteria:

* 1. Age below 40 years and/or onset of symptoms of PAD before the age of 40 years;
* 2. Non-atherosclerotic vascular disease (e.g. Buerger's disease, popliteal entrapment syndrome);
* 3. Limb-threatening (grades III and IV) chronic limb ischemia, manifested by ischemic rest pain, ulceration, or gangrene.
* 4. Patients with a history of malignant or proliferate breast disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Primary: percent change in initial claudication distance (ICD) measured at the 24-week test, compared with that at baseline

SECONDARY OUTCOMES:
Success, defined as an improvement of > 50% in ICD at the 24-week test compared with that at baseline
Percent change in absolute claudication distance (ACD) at the 24-week test, compared with that at baseline,
Functional status / quality of life (QoL) using WIQ and MOS SF-36 questionnaires,
Hemodynamic measurement post treadmill test (ABI/TB).

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (9):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com